CLINICAL TRIAL: NCT00405418
Title: Target Glycemic Control and the Incidence of Documented Symptomatic Hypoglycemia in Insulin naïve Subjects With Type 2 Diabetes Failing on Oral Hypoglycemic Agent(s) and Treated With Insulin Glargine or Insulin Detemir.
Brief Title: Lantus Versus Levemir Treat-To-Target
Acronym: L2T3
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Medical Affairs Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LANTU_C_00579; EUDRACT # : 2006-000324-13
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine; Insulin Detemir

ARMS (2):
- 1 (Experimental): Insulin Glargine
  Interventions: Drug: Insulin glargine
- 2 (Active Comparator): Insulin Detemir
  Interventions: Drug: Insulin Detemir

INTERVENTIONS:
Drug: Insulin glargine — Subcutaneous injection, once a day in the evening
  Arms: 1
Drug: Insulin Detemir — Subcutaneous injection, twice a day at breakfast and before dinner
  Arms: 2

SUMMARY:
Primary objective:

To demonstrate the non-inferiority of insulin glargine in comparison to insulin detemir in term of percentage of patients who reach the target of HbA1c < 7% at the end of the treatment period and do not experience symptomatic hypoglycemia, confirmed by plasma glucose (PG) ≤ 56 mg/dL (3.1 mmol/L)

Secondary objectives:

* To compare between the 2 treatment groups, the percentage of patients who reach the target of HbA1c < 7% and < 6.5% at the end of the treatment period
* To compare the changes in HbA1c and fasting plasma glucose (FPG)
* To compare the evolution of blood glucose profiles
* To compare the day to day FPG variability, the insulin doses
* To determine in each treatment group the biochemical and patient-related determinants of failure to reach HbA1c targets
* To compare the overall incidence and rate of symptomatic hypoglycemia and nocturnal symptomatic hypoglycemia confirmed by PG ≤ 56 mg/dL (3.1 mmol/L)
* To compare over the treatment period, the overall incidence and rate of symptomatic hypoglycemia and symptomatic nocturnal hypoglycemia (with PG ≤ 70 mg/dL [3.9 mmol/L]), of symptomatic day-time hypoglycemia (with PG ≤ 70 mg/dL and with PG ≤ 56 mg/dL), of severe hypoglycemia, of asymptomatic hypoglycemia with PG ≤ 56 mg/dL
* To compare the overall safety: incidence of adverse events (including serious hypoglycemia and local tolerance at injection site), change in body weight, in waist circumference and in waist / hip ratio
* To assess the quality of life and treatment satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes for at least 1 year
* Insulin naïve
* Treated with stable doses of oral antidiabetics for at least 3 months prior to study start, including at least metformin (at least 1g/day)
* 7% ≤ HbA1c ≤ 10.5 %
* Body mass index (BMI) < 40 kg/m²
* Ability and willingness to perform blood glucose monitoring using a blood glucose meter and to use a patient diary

Exclusion Criteria:

* Type 1 diabetes
* Current or previous use of insulin (except for previous treatment of gestational diabetes or brief treatment with insulin for less than 1 week)
* Treatment with glucagon-like peptide (GLP)-1 receptor agonists or with dipeptidyl peptidase (DPP)-IV inhibitors
* Active proliferative diabetic retinopathy, as defined by the application of photocoagulation or surgery, in the 6 months before study entry or any other unstable (rapidly progressing) retinopathy that may require photocoagulation or surgery during the study (an optic fundus examination should have been performed in the 2 years prior to study entry)
* Pregnancy (women of childbearing potential must have a negative pregnancy test at study entry and a medically approved contraceptive method)
* Breast-feeding
* History of hypersensitivity to the study drugs or to drugs with a similar chemical structure
* Treatment with systemic corticosteroids in the 3 months prior to study entry
* Treatment with any investigational product in the 2 months prior to study entry
* Likelihood of requiring treatment during the study period with drugs not permitted by the clinical study protocol
* Clinically relevant cardiovascular, hepatic, neurological, endocrine, or other major disease making implementation of the protocol or interpretation of the study results difficult
* Impaired hepatic function as shown by Alamine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) greater than three times the upper limit of normal range at study entry
* Impaired renal function as shown by serum creatinine ≥ 1.5 mg/dL (≥ 133 μmol/L) in men and ≥ 1.4 mg/dL (124 μmol/L) in women at study entry
* History of drug or alcohol abuse in the last year

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 973 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
HbA1c recorded | At baseline, week 12 and week 24
Self-monitored fasting BG in both treatment arms and pre-dinner BG in detemir arm | On the 4 consecutive days before each visit
Self-monitored BG values from 8-point 24-hour profile recorded on 2 consecutive days | Within the week prior to baseline, week 12 and week 24
Episodes of hypoglycemia (symptomatic, total and categorized as day-time/nocturnal, severe or asymptomatic) | All across the study
Self-monitored BG values whenever patient experiences symptoms possibly related to hypoglycemia. | All across the study

SECONDARY OUTCOMES:
Doses of insulin glargine or insulin detemir | Daily
Laboratory fasting plasma glucose | At baseline, week 12 and week 24
Insulinemia and fasting C-peptide level | At baseline
Lipid profile | at baseline and week 24
Patient reported outcomes (quality of life and treatment satisfaction) | at baseline, week 4, week 12 and at the last visit
Safety data: occurrence of adverse events and weight | assessed at each visit
Waist and hip circumferences | measured at baseline, week 12 and week 24
Systolic and diastolic blood pressure | measured at study entry, baseline, week 12 and week 24
Physical examination | performed at study entry and at last visit.

CONTACTS AND LOCATIONS:
Overall Officials: Valérie Pilorget, Study Director — Sanofi
Locations (20):
- Sanofi-Aventis, North Ryde, Australia
- Sanofi-Aventis, São Paulo, Brazil
- Sanofi-Aventis, Laval, Canada
- Sanofi-Aventis, Hoersholm, Denmark
- Sanofi-Aventis, Helsinki, Finland
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Mumbai, India
- Sanofi-Aventis, Dublin, Ireland
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Porto Salvo, Portugal
- Sanofi-Aventis, Bucharest, Romania
- Sanofi-Aventis, Moscow, Russia
- Sanofi-Aventis, Belgrade, Serbia
- Sanofi-Aventis, Seoul, South Korea
- Sanofi-Aventis, Barcelona, Spain
- Sanofi-Aventis, Stockholm, Sweden
- Sanofi-Aventis, Meyrin, Switzerland
- Sanofi-Aventis, Taipei, Taiwan
- Sanofi-Aventis, Istanbul, Turkey (Türkiye)
- Sanofi-Aventis, Guildford, United Kingdom

REFERENCES:
- [Derived] Swinnen SG, Dain MP, Aronson R, Davies M, Gerstein HC, Pfeiffer AF, Snoek FJ, Devries JH, Hoekstra JB, Holleman F. A 24-week, randomized, treat-to-target trial comparing initiation of insulin glargine once-daily with insulin detemir twice-daily in patients with type 2 diabetes inadequately controlled on oral glucose-lowering drugs. Diabetes Care. 2010 Jun;33(6):1176-8. doi: 10.2337/dc09-2294. Epub 2010 Mar 3. PMID 20200301